CLINICAL TRIAL: NCT05689099
Title: A Study to Demonstrate Bioequivalence Between Semaglutide Drug Product Concentrations 0.68 mg/mL and 1.34 mg/mL
Brief Title: A Research Trial Looking at the Comparability of 2 Different Concentrations of Semaglutide for the 0.5 Milligram (mg) Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-7560; U1111-1280-1368 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2; Healthy Participants
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Participants will be administered a single subcutaneous (s.c.) dose of 0.5 mg semaglutide B (1.34 mg/mL) in Period 1 followed by a single s.c. dose of 0.5 mg semaglutide B (0.68 mg/mL) in Period 2.
  Interventions: Drug: Semaglutide B, 1.34 mg/mL; Drug: Semaglutide B, 0.68 mg/mL
- Sequence B (Experimental): Participants will be administered a single s.c. dose of 0.5 mg semaglutide B (0.68 mg/mL) in Period 1 followed by a single s.c. dose of 0.5 mg semaglutide B (1.34 mg/mL) in Period 2.
  Interventions: Drug: Semaglutide B, 1.34 mg/mL; Drug: Semaglutide B, 0.68 mg/mL

INTERVENTIONS:
Drug: Semaglutide B, 1.34 mg/mL — Participants will receive single dose of 0.5 mg Semaglutide B, 1.34 mg/mL subcutaneously.
Drug: Semaglutide B, 0.68 mg/mL — Participants will receive single dose of 0.5 mg Semaglutide B, 0.68 mg/mL subcutaneously.

SUMMARY:
In this study, a known investigational medicine called 'semaglutide' will be tested in 2 drug concentrations of 0.68 milligram per milliliter (mg/mL) and 1.34 mg/mL. Both drug concentrations are tested for the treatment of type 2 diabetes. The U.S. Food and Drug Administration (FDA), has approved semaglutide in prefilled pen-injector form. Currently, the drug concentration of 1.34 mg/ml can be prescribed in some countries including U.S. The objective of the study is to compare the amount of investigational drug taken up in the body for the 2 drug concentrations. Participants will be divided by chance into 2 groups. Group A will receive a single dose of 0.5 mg semaglutide of the drug concentration 1.34 mg/mL in the first study period; and will receive a single dose of 0.5 mg semaglutide of the drug concentration 0.68 mg/mL in the second study period. Participants assigned to group B will receive the two drug concentrations in the reverse order. Participants will get 1 subcutaneous injection on Day 1 of each of the two study periods. The two injections are separated by 7-11 weeks. The study will last up to approximately 87 to 141 days for each participant. This includes a screening period (up to 4 weeks), study period 1 (5 weeks), washout period (2-6 weeks), and study period 2 (5 weeks). At some periods during the study, participant should not get vaccinations. Participant should agree on timing of vaccination with study doctor. Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 20.0 and 29.9 kilograms per meter square (kg/m^2) (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method
* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, topical medications, highly effective contraceptives and occasional use of paracetamol, ibuprofen and acetylsalicylic acid, within 14 days prior to the day of screening
* Abuse or intake of alcohol, defined as any of the below:

  1. Known or suspected alcohol abuse within 1 year before screening (defined as regular intake of more than an average intake of 24 grams (g) alcohol daily for men and 12 g alcohol daily for women - 12 g of alcohol equals about 300 milliliters (mL) of beer or lager, 100 mL of wine, or 25 mL spirits)
  2. Positive alcohol test at screening
* Abuse or intake of drugs, defined as any of the below:

  1. Known or suspected drug or chemical substance abuse within 1 year before screening
  2. Positive drug of abuse test at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
AUC0-last,sema 0.5mg: Area under the semaglutide concentration time curve from time 0 until last quantifiable measurement after single dose of subcutaneous semaglutide 0.5 mg | 0-840 hours after a single dose of s.c. semaglutide 0.5 mg
  Measured in hours*nanomoles per liter (h*nmol/L).
Cmax,sema,0.5mg: maximum observed semaglutide concentration-time after single dose of subcutaneous semaglutide 0.5 mg administration | 0-840 hours after a single dose of s.c. semaglutide 0.5 mg
  Measured in nanomoles per liter (nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical LA, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com